CLINICAL TRIAL: NCT00590356
Title: A Randomized Comparison of Percutaneous CLip-based Vascular Occluder (Star-Close) Versus Bio-absorble Hemostatic Device (Angio-SEal) for Femoral Artery Hemostasis After Percutaneous Coronary Intervention
Brief Title: Star-Close Versus Angio-Seal for Femoral Artery Hemostasis
Acronym: CLOSE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor, Division of Cardiology, Department of Internal Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20070208
Record Dates: First submitted 2007-12-31; First posted 2008-01-10 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Percutaneous Intervention Via Femoral Artery
Keywords: Device closure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A2 (Active Comparator): AngioSeal®
  Interventions: Device: AngioSeal®
- A1 (Experimental): StarClose®
  Interventions: Device: StarClose®

INTERVENTIONS:
Device: StarClose® — Closure device for femoral artery suture site occlusion
  Other Names: StarClose® vs. AngioSeal®
  Arms: A1
Device: AngioSeal® — Closure device for femoral artery suture site occlusion
  Arms: A2

SUMMARY:
This study was designed to evaluate the efficacy and safety of Starclose (Abbott Vascular Devices) for femoral access site closure in patients undergoing PCI compared to Angio-Seal STS Plus (St. Jude Medical).

DETAILED DESCRIPTION:
The growing success of interventions and requirement for day case or outpatient procedures has led to a concomitant rise in the use of arteriotomy closure devices (ACD) to achieve hemostasis and allow early mobilization following arterial punctures. ACD have emerged as an alternative to traditional mechanical compression after percutaneous coronary intervention (PCI). When compared to manual compression, several studies have confirmed patient comfort, reduced time to achieve hemostasis, reduced time to ambulation, and early discharge.

Recently, CLIP Trial was conducted to evaluated the safety and efficacy of the StarClose device in subjects undergoing diagnostic and interventional catheterization procedures. A total of 17 U.S. sites enrolled 596 subjects, with 483 subjects randomized at a 2:1 ratio to receive StarClose or standard compression of the arteriotomy after the percutaneous procedure. The study included roll-in (n=113), diagnostic (n=208), and interventional (n=275) arms with a primary safety endpoint of major vascular complications through 30 days and a primary efficacy endpoint of postprocedure time to hemostasis. This trial demonstrated that the StarClose Vascular Closure System is noninferior to manual compression with respect to the primary safety endpoint of major vascular events in subjects who undergo percutaneous interventional procedures. StarClose significantly reduced time to hemostasis, ambulation, and dischargeability when compared with compression.

However, there are no studies randomly comparing these two closure devices. Therefore, this study was designed to evaluate the efficacy and safety of Starclose (Abbott Vascular Devices) for femoral access site closure in patients undergoing PCI compared to Angio-Seal STS Plus (St. Jude Medical).

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Patients with appropriate arterial puncture in the common femoral artery eligible for percutaneous closure device deployment Patients undergoing PCI (only 7F sheath)
* Patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Uncontrolled hypertension
* Severe peripheral vascular disease
* Severe femoral artery tortousity and calcification
* Severe obesity (BMI > 35)
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions
* Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
* Patients with cardiogenic shock
* Acute MI patients within symptom onset < 12 hours needing primary angioplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Composite of major vascular complications necessitating surgical or percutaneous repair. | 30-days after randomization

SECONDARY OUTCOMES:
The time to hemostasis. | 30-days after treatment
Procedure time. | 30-days after treatment
Device success. | 30-days after treatment
Procedure success. | 30-days after treatment
Time to ambulation. | 30-days after treatment
Time to discharge. | 30-days after treatment
Subject's comfort level during the deployment of the StarClose using the 11-point Box Scale (BS-11). | 30-days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (1):
- Asan Medical Center, Seoul, South Korea